CLINICAL TRIAL: NCT06156852
Title: A Randomized Clinical Trial Comparing the Effects of Mindfulness-Based Stress Reduction and Cognitive Behavioral Therapy-Based Stress Reduction in Medical Students
Brief Title: Comparing the Effects of Mindfulness-Based and Cognitive Behavioral-Based Stress Reduction in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Aysegul Yay, Research assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GaziU_0001
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Stress; Anxiety; Depressive Symptoms
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction group (MBSR) (Active Comparator): Medical faculty students who volunteered to participate in the study were assessed by a senior psychiatry resident. The students who were found to be eligible to take part in the study were randomized to two groups (MBSR and CBSR groups).
  Interventions: Other: Mindfulness-based stress reduction group
- Cognitive behavioral based stress reduction group (CBSR) (Active Comparator): Medical faculty students who volunteered to participate in the study were assessed by a senior psychiatry resident. The students who were found to be eligible to take part in the study were randomized to two groups (MBSR and CBSR groups).
  Interventions: Other: Cognitive behavioral-based stress reduction group

INTERVENTIONS:
Other: Mindfulness-based stress reduction group — Mindfulness-based stress reduction (MBSR) group interventions were implemented for eight weeks.
  Arms: Mindfulness-based stress reduction group (MBSR)
Other: Cognitive behavioral-based stress reduction group — Cognitive behavioral-based stress reduction group interventions were implemented for eight weeks.
  Arms: Cognitive behavioral based stress reduction group (CBSR)

SUMMARY:
We aimed to compare the effects of the Mindfulness-Based Stress Reduction (MBSR) and the Cognitive Behavioural Stress Reduction (CBSR) group interventions on depression and anxiety symptoms and perceived stress of medical students.

323 medical students applied to participate in one of the group interventions and were assessed with the Mini International Neuropsychiatric Interview. Of these, 253 (77% female, mean age=21.9 ± 2.9 years) were allocated into online MBSR (n=127) and online CBSR (n=126) groups after randomization. Their anxiety and depressive symptoms and perceived stress levels were assessed at baseline and after 8 weeks of interventions.

DETAILED DESCRIPTION:
Objective: Medical students face an enormous amount of stress. They suffer from higher rates of depression, anxiety, and suicide compared to the general population. Despite experiencing more mental health problems, there is a lack of research exploring ways to improve their mental health. Although there are a few small sample studies investigating the effectiveness of Mindfulness-Based Stress Reduction (MBSR) on medical students, there is no study comparing its effectiveness against an active intervention group in the literature.

Aim: We aimed to compare the effects of the Mindfulness-Based Stress Reduction (MBSR) and the Cognitive Behavioural Stress Reduction (CBSR) group interventions on depression and anxiety symptoms and the perceived stress level of medical students.

Methods: The medical students who studied in medical faculties in Ankara/Turkey were asked to participate in our study. In order to invite students to the study, posters announcing our study were put on the boards of the lecture halls of medical faculties, and our posters were shared on social media platforms where these students were involved. After receiving applications from a sufficient number of students who volunteered to participate in the study, the students were assessed online with Mini International Neuropsychiatric Interview by a senior psychiatry resident. Medical students who were eligible to take part in the study were asked to fill out the forms (sociodemographic data form) and scales (Hospital Anxiety-Depression Scale, Perceived Stress Scale) within one week before being allocated into groups. After the students were randomized into two groups with the help of a computer program, stress reduction interventions were conducted for 8 weeks in groups of 10-12 students. After enough participants volunteered to participate in the study, the participants were recruited mainly in two groups and randomized as they were recruited. The first group consisted of 157 participants and the second group consisted of 96 participants. When the group interventions were completed at the end of 8 weeks, the participants were asked to complete the scales (Hospital Anxiety-Depression Scale, Perceived Stress Scale) within one week.

Inclusion Criteria:

* Being a medical student at a university in Ankara
* Being older than 18 years old
* Not having participated in mindfulness-based or cognitive behavioral stress reduction groups or individual therapies
* Volunteering to participate in the study

Exclusion Criteria:

* Having known mindfulness-based stress reduction methods and applied them in their lives
* Having known cognitive behavioral stress reduction methods and applied them in their lives
* Depression and mania severe enough to prevent their participation in the study
* High risk of suicide
* Having a chronic physical condition that may prevent participation in the study
* History of psychotic disorder and/or meeting the diagnosis of psychotic disorder at the assessment stage

Cognitive Behavioral-Based Stress Reduction Groups Stress-coping groups based on cognitive behavioral methods were implemented by adapting them to medical faculty students. The whole intervention was done using the "Zoom" application on the online platform for 8 weeks. Each group meeting was 90 minutes long and held on a specific day and time of the week (19.00-20.30) previously determined by the group members. The groups were planned to consist of 10-12 people and no new members were included after the group started in order not to compromise the integrity of the group.

Mindfulness-Based Stress Reduction Groups Mindfulness-based stress reduction groups consist of structured 8-week 2-hour long group meetings and a 4-hour silence day. Along with mindfulness practices, stress, stress management and use of mindfulness-based practices in daily life and interpersonal communication are the subjects that are being worked on during the sessions. Each group meeting was 120 minutes long and held on a specific day and time of the week (20.00-22.00) previously determined by the group members. The groups were planned to consist of 10-12 people and no new members were included after the group started in order not to compromise the integrity of the group.

Statistical Methods:

SPSS 29 was used for all statistical analysis. In our study, both intention-to-treat (ITT) analysis and per-protocol (PP) analysis were used to assess outcomes. In the ITT analysis, we used multiple imputation to address missing values. All assessments and group interventions were done online. In PP analysis, those who attended five or more sessions were considered to have completed the study. By using two methods and comparing the results of these analyses with each other, we aimed to obtain the most realistic results.

Assessment features-->Statistical methods

Determination of the sample size-->Power analysis(G*power)

Determining the suitability of the data for normal distribution-->Kolmogorov Smirnov / Shapiro-Wilks test Skewness and kurtosis (-1.5- +1.5) Q-Q plot (linearity analysis)

Analyzing the demographic data of the participants-->Percentage distribution, Frequency distribution

Comparison of demographic data of the participants in the two groups-->Chi-square, Independent sample t-test

Comparison of the pre-test and post-test results of the participants in the two groups for each group-->Dependent sample t-test, Mann Whitney U test

Comparison of the change between pre-test and post-test between two groups -->Independent sample t-test, Wilcoxon signed-rank test

Investigate patterns of missingness and assignment of missing data-->Little's test Multiple imputation*

ELIGIBILITY:
Inclusion Criteria:

* Being a medical student at a university in Ankara
* Being older than 18 years old
* Not having participated in mindfulness-based or cognitive behavioral stress reduction groups or individual therapies
* Volunteering to participate in the study

Exclusion Criteria:

* Having known mindfulness-based stress reduction methods and applied them in their lives
* Having known cognitive behavioral stress reduction methods and applied them in their lives
* Depression and mania severe enough to prevent their participation in the study
* High risk of suicide
* Having a chronic physical condition that may prevent participation in the study
* History of psychotic disorder and/or meeting the diagnosis of psychotic disorder at the assessment stage

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Perceived stress level | 8 weeks
  Perceived stress levels were assessed with the Perceived Stress Scale (PSS). This is a widely used scale to assess the effects of different situations on our emotions and perceived stress.
Anxiety level | 8 weeks
  Anxiety symptom levels were assessed with the Hospital anxiety and depression scale (HADS). This scale is a self-assessment scale developed to determine the risk of anxiety and depression in patients with physical illness and primary health care patients and to measure their level and change in severity.
Depressive symptom level | 8 weeks
  Depressive symptom levels were assessed with the Hospital anxiety and depression scale (HADS). This scale is a self-assessment scale developed to determine the risk of anxiety and depression in patients with physical illness and primary health care patients and to measure their level and change in severity.

CONTACTS AND LOCATIONS:
Overall Officials: Selçuk Aslan, MD, Study Director — Gazi University
Locations (1):
- Ayşegül Yay Pençe, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No